CLINICAL TRIAL: NCT01581762
Title: Prospective Comparative Study on Endoscopic Ultrasonography (EUS) - Guided Fine-Needle Aspiration (FNA) Using the 22G Conventional Needles or Procore Needles Without Immediate On-site Cytopathologic Examination
Brief Title: EUS-FNA With 22G Procore Needles vs 22G Conventional Needles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Doctor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ChineseUHK
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Self Efficacy
Keywords: EUS, FNA
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional 22G Needle (Sham Comparator): Device: EUS-FNA with conventional 22G Needle
  Interventions: Procedure: EUS-guided FNA
- 22G Procore Needle (Active Comparator): Device: EUS-FNA with 22G Procore Needle which has a reverse bevel at the tip of the needle to enhance tissue collection
  Interventions: Procedure: EUS-guided FNA

INTERVENTIONS:
Procedure: EUS-guided FNA — EUS-guided FNA with two types of needles - conventional 22G needle (Sham control) and Procore needle (active comparator)
  Other Names: ECHO-HD-22-C, Cook Endoscopy, USA

SUMMARY:
Endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is an important investigation tool to obtain tissue for diagnosis. Nowadays, the performance of EUS-FNA varies with accuracy rates ranging from 60% - 100%. Needles with different diameters have been explored to retrieve tissue specimens. The diagnostic yields, successful rates and safety profiles are similar. It has been suggested that although thinner needles provide less cellular material than do larger needles, the specimens from the former are less contaminated by blood, and thus easier to interpret. In addition, thinner needles may be easier to use because of greater flexibility, particularly for locations requiring important scope bending. As a result, a new 22G FNA needle has been designed in order to improve the tissue-sampling rate (ECHO-HD-22-C, Cook Endoscopy, USA). There is a reverse bevel at the tip of the new needle with promotes collection of core sample by shearing material from target lesion during retrograde movement of the needle in the lesion. The feasibility and safety of this newly design EUS-FNA needle have been demonstrated in a recent multicenter, pooled, cohort study using the 19G version. Successful puncture was technically feasible in 98.2% of cases and the overall accuracy of 92.9%. There were no complications related to the technique.

The aim of this study is to compare the tissue-sampling rate and the diagnostic accuracy rate of EUS-FNA between the uses of the convention and newly designed 22-gauge needles.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) - guided fine needle aspiration (FNA) is a well-established technique for tissue sampling of intestinal and extra-intestinal mass lesions. The accuracy of EUS-guided FNA varies from 60% - 100% with a complication rate of 0% - 3%. The diagnostic accuracy of the procedure can be improved by the use immunohistochemical studies and genetic analyses.It may also be improved by obtaining a larger biopsy specimen with a core biopsy needle. However, puncturing with a core-biopsy needle may not be always feasible due to the technical difficulty of inserting the larger needle through the bended endoscope. As a result, the advantage of a core-biopsy needle on providing a larger amount of cellular material is offset by a higher rate of technical failures, especially in the setting of a transduodenal puncture. Recently, a new 22G FNA needle with a reverse bevel at the tip has become available (ECHO-HD-22-C, Cook Endoscopy, USA.). The design of the device promotes the collection of core samples by shearing material from target lesion during retrograde movement of the needle in the lesion. Hence, the aim of this study is to compare the tissue-sampling rate and the diagnostic accuracy rate of EUS-FNA using 22G conventional and Procore needles.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-80 undergoing EUS-guided tissue acquisition
* Informed consent available

Exclusion Criteria:

* Coagulopathy
* Previous history of upper gastrointestinal surgery
* Contraindications for conscious sedation
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with cyto-histopathology confirmed neoplasms diagnosed by EUS-guided FNA | 1 year
  A positive diagnosis of malignancy by an EUS biopsy specimen is accepted as a true positive. A benign diagnosis is confirmed by surgical tissue samples when available or clinical follow-up after 1 year.

SECONDARY OUTCOMES:
Diagnostic accuracy | 1 year
  A positive diagnosis of malignancy by an EUS biopsy specimen is accepted as a true positive. A benign diagnosis is confirmed by surgical tissue samples when available or clinical follow-up after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: CHARING C CHONG, MBChB, Principal Investigator — Department of Surgery, CUHK
Locations (1):
- Department of Surgery, Hong Kong, Hong Kong

REFERENCES:
- [Background] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Background] Kida M. Pancreatic masses. Gastrointest Endosc. 2009 Feb;69(2 Suppl):S102-9. doi: 10.1016/j.gie.2008.12.010. No abstract available. PMID 19179132
- [Background] Gress F, Gottlieb K, Sherman S, Lehman G. Endoscopic ultrasonography-guided fine-needle aspiration biopsy of suspected pancreatic cancer. Ann Intern Med. 2001 Mar 20;134(6):459-64. doi: 10.7326/0003-4819-134-6-200103200-00010. PMID 11255521
- [Background] O'Toole D, Palazzo L, Arotcarena R, Dancour A, Aubert A, Hammel P, Amaris J, Ruszniewski P. Assessment of complications of EUS-guided fine-needle aspiration. Gastrointest Endosc. 2001 Apr;53(4):470-4. doi: 10.1067/mge.2001.112839. PMID 11275888
- [Background] Yusuf TE, Ho S, Pavey DA, Michael H, Gress FG. Retrospective analysis of the utility of endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) in pancreatic masses, using a 22-gauge or 25-gauge needle system: a multicenter experience. Endoscopy. 2009 May;41(5):445-8. doi: 10.1055/s-0029-1214643. Epub 2009 May 5. PMID 19418399
- [Background] Itoi T, Itokawa F, Kurihara T, Sofuni A, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Kawai T, Moriyasu F. Experimental endoscopy: objective evaluation of EUS needles. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):509-16. doi: 10.1016/j.gie.2008.07.017. PMID 19231491
- [Background] Yun SS, Remotti H, Vazquez MF, Crapanzano JP, Saqi A. Endoscopic ultrasound-guided biopsies of pancreatic masses: comparison between fine needle aspirations and needle core biopsies. Diagn Cytopathol. 2007 May;35(5):276-82. doi: 10.1002/dc.20621. PMID 17427217
- [Background] Fritscher-Ravens A, Topalidis T, Bobrowski C, Krause C, Thonke E, Jackle S, Soehendra N. Endoscopic ultrasound-guided fine-needle aspiration in focal pancreatic lesions: a prospective intraindividual comparison of two needle assemblies. Endoscopy. 2001 Jun;33(6):484-90. doi: 10.1055/s-2001-14970. PMID 11437040
- [Background] Savides TJ, Donohue M, Hunt G, Al-Haddad M, Aslanian H, Ben-Menachem T, Chen VK, Coyle W, Deutsch J, DeWitt J, Dhawan M, Eckardt A, Eloubeidi M, Esker A, Gordon SR, Gress F, Ikenberry S, Joyce AM, Klapman J, Lo S, Maluf-Filho F, Nickl N, Singh V, Wills J, Behling C. EUS-guided FNA diagnostic yield of malignancy in solid pancreatic masses: a benchmark for quality performance measurement. Gastrointest Endosc. 2007 Aug;66(2):277-82. doi: 10.1016/j.gie.2007.01.017. PMID 17643700
- [Background] Harewood GC, Wiersema MJ. Endosonography-guided fine needle aspiration biopsy in the evaluation of pancreatic masses. Am J Gastroenterol. 2002 Jun;97(6):1386-91. doi: 10.1111/j.1572-0241.2002.05777.x. PMID 12094855
- [Background] Eloubeidi MA, Chen VK, Eltoum IA, Jhala D, Chhieng DC, Jhala N, Vickers SM, Wilcox CM. Endoscopic ultrasound-guided fine needle aspiration biopsy of patients with suspected pancreatic cancer: diagnostic accuracy and acute and 30-day complications. Am J Gastroenterol. 2003 Dec;98(12):2663-8. doi: 10.1111/j.1572-0241.2003.08666.x. PMID 14687813